CLINICAL TRIAL: NCT00296491
Title: A Multicenter, Randomized, Double-Blind, Triple-Dummy, Placebo-Controlled, Parallel Group, Four-Week Study Assessing the Efficacy of Fluticasone Propionate Aqueous Nasal Spray 200mcg QD Versus Montelukast 10mg QD in Adolescent and Adult Subjects With Asthma and Seasonal Allergic Rhinitis Who Are Receiving ADVAIR DISKUS® 100/50mcg BID or Placebo BID
Brief Title: Study Of Allergic Rhinitis In Patients Who Also Have Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA103575
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Fluticasone; Salmeterol Xinafoate; montelukast; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) (Active Comparator): Fluticasone propionate/salmeterol DISKUS combination product (FSC) twice daily (BID) plus vehicle placebo nasal spray once daily (QD) plus montelukast capsule 10mg (MON) QD
  Interventions: Drug: fluticasone propionate/salmeterol (FSC); Drug: montelukast (MON); Drug: placebo nasal; Drug: ADVAIR DISKUS
- Fluticasone Propionate/Salmeterol (FSC) (Active Comparator): FSC BID plus vehicle placebo nasal spray QD plus placebo capsule QD
  Interventions: Drug: fluticasone propionate/salmeterol (FSC); Drug: placebo nasal; Drug: ADVAIR DISKUS; Drug: placebo capsule
- Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) (Active Comparator): Fluticasone propionate/salmeterol DISKUS combination product (FSC)100/50mcg BID plus fluticasone propionate aqueous nasal spray 200mcg (FPANS) QD plus placebo capsule QD
  Interventions: Drug: fluticasone propionate/salmeterol (FSC); Drug: fluticasone propionate (FP); Drug: ADVAIR DISKUS; Drug: placebo capsule
- Montelukast (MON) (Active Comparator): Placebo DISKUS BID plus vehicle placebo nasal spray QD plus MON QD
  Interventions: Drug: montelukast (MON); Drug: placebo nasal; Drug: placebo DISKUS

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol (FSC) — fluticasone propionate/salmeterol DISKUS combination
  Arms: Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS); Fluticasone Propionate/Salmeterol (FSC); Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON)
Drug: montelukast (MON) — montelukast capsule
  Arms: Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON); Montelukast (MON)
Drug: fluticasone propionate (FP) — fluticasone propionate aqueous nasal spray
  Arms: Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS)
Drug: placebo nasal — vehicle placebo nasal spray
  Arms: Fluticasone Propionate/Salmeterol (FSC); Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON); Montelukast (MON)
Drug: ADVAIR DISKUS — ADVAIR DISKUS
  Arms: Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS); Fluticasone Propionate/Salmeterol (FSC); Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON)
Drug: placebo capsule — placebo capsule
  Arms: Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS); Fluticasone Propionate/Salmeterol (FSC)
Drug: placebo DISKUS — placebo DISKUS
  Arms: Montelukast (MON)

SUMMARY:
This study will last up to 6 weeks. Subjects will visit the clinic up to 5 times. Certain clinic visits will include a physical examination, medical history review, and lung function tests. All study related medications and medical examinations will be provided at no cost to the subject. The drugs used in this study are approved for the age group under study.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Triple-Dummy, Placebo-Controlled, Parallel Group, Four-Week Study Assessing the Efficacy of Fluticasone Propionate Aqueous Nasal Spray 200mcg QD versus Montelukast 10mg QD in Adolescent and Adult Subjects with Asthma and Seasonal Allergic Rhinitis Who are Receiving ADVAIR DISKUS® 100/50mcg BID or Placebo BID

ELIGIBILITY:
INCLUSION CRITERIA:

A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:

* Consent: A signed and dated written informed consent must be obtained from the subject or subject's legally acceptable representative prior to study participation. An informed consent must be signed prior to any change in the subject's medication regimen, including withholding medications prior to Visit 1.
* Gender: Male or female. Females are eligible to participate only if they are currently not pregnant and not lactating. Females of child-bearing potential will be required to use a highly effective method for avoiding pregnancy (i.e., contraception with a failure rate of <1% per year). Female subjects of child-bearing potential will undergo a urine pregnancy test at Visits 1, 2, 3, and 4. Any female who becomes pregnant during the study will be withdrawn. Female subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* Age: 15 years and older.
* Asthma Diagnosis: A diagnosis of persistent asthma, for at least three months, as defined by the following American Thoracic Society definition:

Asthma is a clinical syndrome characterized by increased responsiveness of the tracheobronchial tree to a variety of stimuli. The major symptoms of asthma are paroxysms of dyspnea, wheezing, and cough, which may vary from mild and almost undetectable to severe and unremitting (status asthmaticus). The primary physiological manifestation of this hyperresponsiveness is variable airway obstruction. This can take the form of spontaneous fluctuations in the severity of obstruction, substantial improvements in the severity of obstruction following bronchodilators or corticosteroids, or increased obstruction caused by drugs or other stimuli [American Thoracic Society, 1987a].

NOTE: Intermittent and seasonal asthma, as well as exercise-induced bronchospasm alone, are excluded.

* Asthma Therapy: 3 months' prior and current use of one of the following asthma therapies, with no change in regimen during the month prior to Visit 1:

  * Scheduled or as-needed inhaled or oral short-acting beta2-agonist (SABA). Subjects must be able to replace their current short-acting beta2-agonist with albuterol/salbutamol, to be used only on an as-needed basis for the duration of the study.
  * Allowed non-corticosteroid controller therapy (e.g., anticholinergics and cromolyn).
  * One of the following inhaled corticosteroids taken at the corresponding daily dose:

criteria.

Inhaled Corticosteroid (Total Daily Dose) Beclomethasone dipropionate (≤420mcg) Beclomethasone dipropionate HFA (≤240mcg) Budesonide (≤400mcg) Flunisolide (≤1000mcg) Fluticasone propionate inhalation aerosol (≤220mcg) Fluticasone propionate inhalation powder (≤250mcg) Mometasone furoate (≤220mcg) Triamcinolone acetonide (≤1000mcg) Subjects taking ADVAIR 100/50mcg BID are eligible to replace ADVAIR with FLOVENT HFA 110mcg BID for 14 days prior to Visit 1. This change will be at the Investigator's clinical discretion, taking each individual's current and past asthma stability into account. The subject must be aware of the risks and benefits of switching their medication and acknowledge this by signing an informed consent prior to any change in the subject's medication regimen.

* Asthma Severity: An FEV1 between 65% - 95% of predicted value at Visit 1 after withholding asthma medications as detailed in the protocol.

At Visit 2, subjects must also be experiencing minimum asthma symptoms as defined in Section 5.2.3, "Randomization Criteria", and in Section 6.2 of the protocol.

Predicted FEV1 will be based on the National Health and Nutrition Examination Survey (NHANES III) predicted normal values [Hankinson, 1999].

* Rhinitis Diagnosis: A diagnosis of seasonal allergic rhinitis defined as follows:

  * A clinical history (written or verbal confirmation) of allergic rhinitis with the seasonal onset and offset of nasal allergy symptoms during each of the previous 2 relevant allergy seasons (captured in source documents only).

AND •A positive skin test reaction to a geographically relevant seasonal allergen, as determined by the skin prick method, within 24 months prior to or at Visit 1.

For the purposes of this study, a positive skin test reaction is defined as a wheal diameter that is at least 3mm greater than diluent control using 1:20 W:V glycerinated solution.

•At Visit 2, subjects must also be experiencing minimum rhinitis symptoms as defined in Section 5.2.3, "Randomization Criteria", and in Section 6.2 of the protocol.

* Geographical Location: Active residence within a geographical region where exposure to a relevant seasonal allergen is expected to be significant during the entire study period.

Note: The principal investigator is responsible for tracking and recording pollen counts for geographically relevant seasonal allergens throughout the entire study. Alternatively, this information may be obtained from a reputable source from within the same geographical area.

EXCLUSION CRITERIA:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Currently Diagnosed with Life-Threatening Asthma: An episode or episodes of asthma requiring intubation associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* Asthma Instability: Hospitalization for asthma within 6 months of Visit 1.
* Concurrent Respiratory Disease: Current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, emphysema, or any other respiratory abnormalities other than asthma.
* Nasal Obstruction: Severe physical obstruction of the nose (e.g., deviated septum) that could affect the deposition of double-blind intranasal study drug.
* Nasal History: History of nasal septal perforation or recent nasal septal surgery.
* Other Concurrent Conditions/Diseases: Any evidence of rhinitis medicamentosa, history of glaucoma and/or cataracts or ocular herpes simplex, or any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study.

The list of additional excluded conditions/diseases includes, but is not limited to: cardiac arrhythmias; congestive heart failure; coronary artery disease; poorly controlled diabetes, poorly controlled hypertension, poorly controlled peptic ulcer, hematologic, hepatic, or renal disease; immunologic compromise; current malignancy; current or quiescent tuberculosis, and Cushing's or Addison's disease.

* Drug Allergy: Any immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, leukotriene modifier, or any intranasal, inhaled, or systemic corticosteroid therapy, or sensitivity to aspirin or other NSAIDS. Subjects with severe milk protein allergies are also excluded from participation.
* Respiratory Tract Infections: Any sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection that has not resolved at least 14 days immediately preceding Visit 1, or for which antibiotic therapy has not been completed at least 14 days prior to Visit 1.
* Concurrent Medications: Concurrent use of any of the following medications that may affect the course of asthma, rhinitis, or interact with sympathomimetic amines or montelukast.

  * Beta-blockers
  * tricyclic antidepressants
  * monoamine oxidase inhibitors
  * phenobarbital
  * rifampin
  * ritonavir
  * ketoconazole
* Systemic Corticosteroids: Use of oral or parenteral systemic corticosteroids within 28 days of Visit 1, or requirement for more than two courses of parenteral systemic corticosteroids for asthma within 6 months of Visit 1.

NOTE: Topical hydrocortisone cream or ointment (1% or less) is permitted during the study.

* Excluded Rhinitis Medications: The following rhinitis medications must be withheld during the corresponding "exclusion period" prior to Visit 1 and are not allowed any time during the study, unless dispensed as double-blind study drug:

Medication (Exclusion Period Prior to Visit 1) Intranasal and ocular corticosteroids (28 days) Leukotriene modifiers (e.g., Singulair, Accolate, Zyflo) (28 days) Intranasal and ocular cromolyn (14 days) Long-acting antihistamines (e.g., loratadine, cetirizine) (10 days) Short-acting antihistamines (includes prescription and OTC) (72 hours) Oral and intranasal decongestants (72 hours) Intranasal anticholinergics (e.g., Atrovent) (24 hours)

* Excluded Asthma Medications: The following asthma medications must be withheld during the corresponding "exclusion period" prior to Visit 1.

These asthma medications, with the exception of an inhaled corticosteroid/long-acting beta2-agonist combination product and Xolair, may be continued during the run-in period of the study (between Visits 1 and 2), but must be withheld prior to Visit 2 for the appropriate "exclusion period" as shown below.

These asthma medications are not allowed any time after randomization at Visit 2 (with the exception of as as-needed rescue albuterol/salbutamol), unless dispensed as double-blind study drug:

Medicationª (Exclusion Period Prior to Visit 1 and/or Visit 2) Inhaled corticosteroid/long-acting beta2-agonist combination product (e.g., ADVAIR) (14 days) Inhaled anticholinergics (e.g., Atrovent, Combivent, Spiriva) (24 hours) Theophylline products (48 hours) Inhaled cromolyn or nedocromil (24 hours) Inhaled corticosteroids (12 hours) Long-acting beta2-agonists (e.g., Foradil, SEREVENT™) (14 days) Oral beta2-agonists (12 hours) Inhaled short-acting beta2-agonists^b (e.g., Proventil) (6 hours) Xolair (12 months)

1. For the leukotriene modifier "exclusion period" prior to Visit 1, refer to Exclusion Criterion 11.
2. Replaced at Visit 1 with albuterol/salbutamol.

   * Ophthalmic preparations: Use of artificial tears, eyewashes, homeopathic preparations, irrigation solutions, lubricants, sympathomimetic preparations, vasoconstrictors, or combinations of any of the aforementioned products during the study.
   * Immunosuppressive Medications: Use of immunosuppressive medications during the study.

NOTE: Immunotherapy for the treatment of allergies is allowed during the study, provided that it was not initiated within 30 days of Visit 1, the dose has remained fixed over the 30 days prior to Visit 1, and the dose will remain fixed for the duration of the study.

* Positive Pregnancy Test: A positive pregnancy test at Visit 1.
* Tobacco Use: Greater than a 10 pack-year history of cigarette smoking or use of any tobacco products within 1 year of Visit 1. This includes cigarettes, cigars, pipe, chewing tobacco, and snuff.

Note: Pack years = number of cigarettes smoked per day divided by 20, multiplied by the number of years of smoking.

* Questionable Validity of Consent: Any infirmity or disability that would limit the subject's consent or geographic location that would limit the compliance for scheduled visits.
* Investigational Medications: Use of any investigational drug within 30 days of Visit 1.
* 3rd shift/Nighttime employment: Any employment during the nighttime hours (10 p.m. - 6 a.m.) or 3rd shift.
* Site affiliation: Participation of anyone associated with the administration of the study or their immediate family members

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (91):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, North Andover, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Forked River, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Parma, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Savannah, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Kirkland, Washington
- Canada (10):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kanata, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Niagara Falls, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Katial RK, Oppenheimer JJ, Ostrom NK, Mosnaim GS, Yancey SW, Waitkus-Edwards KR, Prillaman BA, Ortega HG. Adding montelukast to fluticasone propionate/salmeterol for control of asthma and seasonal allergic rhinitis. Allergy Asthma Proc. 2010 Jan-Feb;31(1):68-75. doi: 10.2500/aap.2010.31.3306. PMID 20167147
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADA103575 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Flut Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS): Flut Prop = Fluticasone Propionate.
Period: Overall Study
Arm/Group | Flut Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC) | Montelukast (MON)
Started | 182 (Please note: Outcome Measures generally conducts analysis of 2 of the 4 Arms at a time.) | 182 | 180 | 181
Completed | 140 | 129 | 137 | 138
Not Completed | 42 | 53 | 43 | 43
Not completed — Low Pollen Counts | 18 | 26 | 25 | 16
Not completed — Protocol Violation | 4 | 6 | 2 | 3
Not completed — Adverse Event | 1 | 3 | 1 | 4
Not completed — Withdrawn due to Asthma | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 7 | 3 | 3 | 2
Not completed — Non-Compliance | 12 | 13 | 10 | 14
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON): Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) = FSC twice a day (BID), plus vehicle placebo nasal spray once a day (QD), plus MON once a day (QD)
- Fluticasone Propionate/Salmeterol (FSC): Fluticasone Propionate/Salmeterol (FSC) = FSC BID, plus vehicle placebo nasal spray once a day (QD), plus placebo capsule once a day (QD).
- Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS): Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) = FSC twice a day (BID), plus FPANS (once a day) QD, plus placebo capsule once a day (QD).
- Montelukast (MON): Montelukast (MON) = Placebo DISKUS BID, plus vehicle placebo nasal spray once a day (QD), plus MON (once a day) QD.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC) | Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) | Montelukast (MON) | Total
Number analyzed (Participants) | 182 | 180 | 182 | 181 | 725
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (13.54) | 34.5 (14.64) | 34.9 (12.62) | 34.5 (12.47) | 34.2 (13.34)
Gender [Count of Participants; unit: Participants]
  Female | 115 | 102 | 120 | 112 | 449
  Male | 67 | 78 | 62 | 69 | 276
Race/Ethnicity, Customized [Number; unit: participants]
  White | 138 | 138 | 143 | 145 | 564
  African American/African Heritage | 34 | 35 | 31 | 30 | 130
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 9 | 5 | 5 | 5 | 24
  Native Hawaiian or other Pacific Islander | 1 | 1 | 1 | 1 | 4
  Unknown | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at Endpoint in Morning Peak Expiration Flow (PEF) for Intent-to-Treat Population
Description: Endpoint was defined as the average of the data reported from the last week of treatment. Data collected by patient throughout the treatment period between visits. The peak expiratory flow rate measures how fast a person can breathe out (exhale) air. It is one of many tests that measure how well your airways work.
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: The Intent-to-Treat (ITT) population, the basis for superiority comparisons between FSC and MON in the context of asthma measures, included all subjects randomized to double-blind treatment.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Fluticasone Prop/Salmeterol (FSC) | Montelukast (MON)
Number analyzed (Participants) | 179 | 181
L/min | 26.4 (4.10) | 3.6 (3.28)
Statistical Analysis 1: Comparison: Fluticasone Prop/Salmeterol (FSC) vs Montelukast (MON); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 23.2, 95% CI [12.5 to 33.8], Standard Error of Mean 5.41 — Treatment Difference = FSC - MON

2. Primary Outcome: Mean Change From Baseline at Endpoint in Morning Peak Expiratory Flow (PEF) for Per Protocol Population
Description: as for outcome 1
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: The Per Protocol population, the basis for equivalence comparison between FSC and FSC+MON in terms of asthma measures, included subjects from the ITT population who did not deviate significantly from the protocol.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Flut Prop/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 83 | 88
L/min | 30.9 (4.92) | 35.2 (6.41)
Statistical Analysis 1: Comparison: Flut Prop/Salmeterol/Montelukast (FSC+MON) vs Fluticasone Propionate/Salmeterol (FSC); Test type: Non-Inferiority or Equivalence — Given estimates, and assuming a significance level of a=0.05, a sample size of 133 subjects per treatment was determined to be sufficient to provide 80% power to show equivalance; p < 0.127, t-test, 2 sided; Mean Difference (Net) = -8.9, 95% CI [-24.6 to 6.9], Standard Error of Mean 8.00 — Treatment Difference=FSC+MON-FSC

3. Secondary Outcome: Rhinitis: Mean Change From Baseline at 1-2 Weeks in Daytime Total Nasal Symptom Scores (D-TNNS).
Description: The sum of scores of each of the four daytime symptoms (nasal congestion, itching, rhinorrhea, and sneezing). Scale: 0=none (no sign/symptom evident)1=mild (sign/symptom clearly present; easily tolerated)2=moderate (definite awareness of sign/symptom that is bothersome but tolerable)3=severe (sign/symptom is hard to tolerate)
Time Frame: Baseline to 1-2 Weeks
Population: The Intent-to-Treat (ITT) population, the basis for superiority comparisons between FSC+FPANS and FSC+MON in the context of rhinitis measures, included all subjects randomized to double-blind treatment. Families of secondary efficacy measures were each adjusted for multiplicity using Hochberg's method.
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Fluticasone Prop/Salmeterol/Montelukast (FSC+MON) | Fluticasone Prop/Salmeterol/Flut Nasal Spray (FSC+FPANS)
Number analyzed (Participants) | 181 | 181
Points on a Scale | -2.3 (0.16) | -3.0 (0.18)

4. Secondary Outcome: Rhinitis: Mean Change From Baseline at 1-2 Weeks in Nightime Total Nasal Symptom Scores (N-TNSS)
Description: The scores of 3 nighttime symptoms (nasal congestion upon awakening, difficulty going to sleep due to nasal symptoms, nighttime awakenings due to nasal symptoms). Scale: 0=not noticeable, 1=noticeable but not bothersome, 2=noticeable and bothersome some of the time, 3=bothersome most of the time and/or very bothersome some of the time.
Time Frame: Baseline To 1-2 Weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Flut Prop/Salmeterol/Flut Nasal Spray (FSC+FPANS) | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON)
Number analyzed (Participants) | 181 | 181
Points on a Scale | -2.0 (0.13) | 1.7 (0.13)

5. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Predose Morning Forced Expiratory Volume (FEV1) for Intent-to-Treat Population
Description: Endpoint was defined as the average of the last week's worth of evaluable data. The volume of air that can be forced out taking a deep breath, an important measure of pulmonary function. FEV1 is forced expiratory volume in one second.
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: The Intent-to-Treat (ITT) population, the basis for superiority comparisons between FSC and MON in the context of asthma measures, included all subjects randomized to double-blind treatment. Families of secondary efficacy measures were each adjusted for multiplicity using Hochberg's method.
Measure: Mean (Standard Error); unit: L/sec
Arm/Group | Fluticasone Propionate/Salmeterol (FSC) | Montelukast (MON)
Number analyzed (Participants) | 178 | 180
L/sec | 0.15 (0.02) | 0.04 (0.03)

6. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Predose Morning Forced Expiratory Volume (FEV1) for Per Protocol Population
Description: as for outcome 5
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: The Per Protocol population, the basis for equivalence comparison between FSC and FSC+MON in terms of asthma measures, included subjects from the ITT population who did not deviate significantly from the protocol. Families of secondary efficacy measures were each adjusted for multiplicity using Hochberg's method.
Measure: Mean (Standard Error); unit: L/sec
Arm/Group | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 83 | 88
L/sec | 0.27 (0.04) | 0.13 (0.04)

7. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Percentage of Asthma Symptom-Free Days for Intent-to-Treat Population
Description: Endpoint was defined as the average of the data reported from the last week of treatment.Asthma symptom scores and the subject-rated overall satisfaction with treatment, related to the percentage of asthma symptom-free days. Same scale used as in outcome 8.
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage of asthma symptom-free days
Arm/Group | Fluticasone Propionate/Salmeterol (FSC) | Montelukast (MON)
Number analyzed (Participants) | 179 | 181
Percentage of asthma symptom-free days | 34.8 (2.94) | 26.1 (2.83)

8. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Percentage of Asthma Symptom-Free Days for Per Protocol Population
Description: Asthma symptom score:0=no symptoms,1=symptoms 1 short period,2=symptoms 2 or more short periods,3=symptoms most of day not affect activities,4=symptoms most of day did affect activities,5=symptoms severe.Overall satisfaction score:0=very dissatisfied,1=dissatisfied,2=slightly dissatisfied,3=neutral,4=slightly satisfied,5=satisfied 6=very satisfied
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Percentage of asthma symptom-free days
Arm/Group | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 83 | 88
Percentage of asthma symptom-free days | 34.8 (4.32) | 37.1 (4.23)

9. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Percentage of Albuterol-Salbutamol Free Days for Intent-to-Treat Population
Description: Endpoint was defined as the average of the data reported from the last week of treatment. Albuterol/salbutamol use (related to percentage of asthma rescue-free days).
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage of rescue-free days
Arm/Group | Fluticasone Propionate/Salmeterol (FSC) | Montelukast (MON)
Number analyzed (Participants) | 179 | 181
Percentage of rescue-free days | 37.5 (2.84) | 26.7 (2.92)

10. Secondary Outcome: Asthma: Mean Change From Baseline at Endpoint in Percentage of Albuterol/Salbutamol-Free Days for Per Protocol Population
Description: as for outcome 9
Time Frame: Baseline to Endpoint (weeks 3-4)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Percentage of rescue-free days
Arm/Group | Fluticasone Propionate + Salmeterol & Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 83 | 88
Percentage of rescue-free days | 41.2 (3.97) | 42.9 (4.20)

ADVERSE EVENTS:
Arm/Group | Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) | Fluticasone Propionate/Salmeterol (FSC) | Montelukast (MON)
Serious Adverse Events (participants affected / at risk) | 0/182 | 1/182 | 1/180 | 1/181
Other Adverse Events (participants affected / at risk) | 32/182 | 32/182 | 42/180 | 41/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) (N=182) | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) (N=182) | Fluticasone Propionate/Salmeterol (FSC) (N=180) | Montelukast (MON) (N=181)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Prop/Salmeterol/Flut Prop Nasal Spray (FSC+FPANS) (N=182) | Fluticasone Propionate/Salmeterol/Montelukast (FSC+MON) (N=182) | Fluticasone Propionate/Salmeterol (FSC) (N=180) | Montelukast (MON) (N=181)
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 4
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 4 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 7 | 7 | 8 | 8
Sinus headache (Nervous system disorders) | 0 | 2 | 3 | 1
Migraine (Nervous system disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 3
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Chest pain (General disorders) | 0 | 1 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1
Eye pruritis (Eye disorders) | 2 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Anorgasmia (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.